CLINICAL TRIAL: NCT02736006
Title: Decreases in Diffusing Lung Capacity for Carbon Monoxide (DLCO) in Occupational Divers and Their Impact on Decompression Sickness Risks
Acronym: DACODEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RB15.173 (DACODEC)
Record Dates: First submitted 2016-03-16; First posted 2016-04-13 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Decompression Sickness
Keywords: Alveolo-capillar membrane; decompression illness; diving; occupational
MeSH Terms: conditions — Decompression Sickness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 20 meters air dive (Experimental)
  Interventions: Other: 20 meters air dive

INTERVENTIONS:
Other: 20 meters air dive — A dive in the depth of 20 m during 40 minutes. The divers will be evaluated before and 30, 60, 180 minutes after a 20 meters air dive. Venous bubbles will be detected by precordial Doppler 30 minutes after the dive.
  In association with this Doppler, Flow Mediated Dilation, blood samples analysing inflammatory and thrombotic factors and other biomarkers will be explored before and after the dive in order to know how vascular and respiratory tracts in this environment react.

SUMMARY:
Diving disorders and particularly Decompression sickness (DCS) represent a major concern in recreational and occupational pressure-related activities. As a result of decompression from higher to lower ambient pressure bubbles which are formed in vascular flow and in tissues take part in embolism then resulting in DCS. Individual factors such as vascular or respiratory defects are now considered to increase the risk of this dysbarism disease.

DETAILED DESCRIPTION:
2 groups of occupational divers will be separated after a fitness medical examination by regarding DLCO decrease or not.

The divers will be evaluated before and 30, 60, 180 minutes after a 20 meters air dive. Venous bubbles will be detected by precordial Doppler 30 minutes after the dive.

In association with this Doppler, Flow Mediated Dilation, blood samples analysing inflammatory and thrombotic factors and other biomarkers will be explored before and after the dive in order to know how vascular and respiratory tracts in this environment react.

ELIGIBILITY:
Inclusion Criteria:

* Be professional and voluntary diver
* Man or woman aged 18 years or older
* Diffusing Lung Capacity for Carbon Monoxide measured beforehand in the study
* No medical contraindication for hyperbaric
* No hyperbaric constraint in 3 days before the dive
* No prior Decompression sickness
* Not to follow medicinal treatment modifying the vascular endothelial and/or the coagulation and/or the respiratory function
* Patient affiliated to social security
* Informed and signed

Exclusion Criteria:

* Concomitant pathology identified by the Investigator, justifying a contraindication for hyperbaric
* Pregnant and nursing mothers
* Patient who refuse to sign consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-03-22 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
Venous bubbles will be detected by precordial Doppler | 30 minutes after the dive
  Venous bubbles will be detected by precordial Doppler

SECONDARY OUTCOMES:
Vascular abnormality | 60 minutes after the dive
  Assessement of microvascular reactivity by brachial artery flow mediated dilation
Coagulation activation | 60 minutes after the dive
  Assessment of blood coagulation factor after the dive
Inflammatory activation | 60 minutes after the dive
  Assessment of inflammatory factor after the dive

CONTACTS AND LOCATIONS:
Locations (1):
- Brest, University Hospital, Brest, France